## **Protocol**

# PROTOCOL NUMBER: EC22-008

## **STUDY TITLE:**

A Real World Evidence Study of Danish Fabry patients: a > 20-year Longitudinal Retrospective Analysis of Prospectively Collected Data.

VERSION: 1.0 (Original) DATE: 30 June 2023

#### **SPONSOR:**

Amicus Therapeutics Ltd.
One Globeside, Fieldhouse Ln, Marlow SL7 1HZ, UK

## **Study information**

| Title | Real World Evidence study of Danish Fabry patients: a >20-year longitudinal retrospective analysis of prospectively collected data. |
|---|---|
| Protocol version identifier | V1 |
| Date of last version of protocol | |
| Active substance | NA |
| Medicinal product | NA |
| Product reference | NA |
| Procedure number | |
| Marketing authorisation holder(s) | |
| Joint PASS | |
| MAH(s) contact | |
| Research question and objectives | Research Question |
| | Is the incidence and prevalence of Fabry associated clinical events (FACEs) (cardiac, renal and cerebrovascular) associated with sex, genotype, phenotype at time of diagnosis, biomarkers, and Fabry specific therapy? |
| | Objectives |
| | To investigate time to first Fabry associated clinical events (FACEs) (cardiac, renal, and cerebrovascular) with particular focus on Migalastat clinical outcomes and treatment outcomes preceding Migalastat therapy. |
| | To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment. |
| | To describe FACEs in accordance with different genoand phenotypic groups. |
| | To investigate the incidence and time to a first fatal or non-fatal cardiac, renal and cerebrovascular clinical event, separated by each category. |

| Title | Real World Evidence study of Danish Fabry patients: a >20-year longitudinal retrospective analysis of prospectively collected data. |
|---|---|
| | Primary objectives |
| | To investigate time to first Fabry associated clinical events (FACE) (cardiac, renal, and cerebrovascular) with particular focus on Migalastat clinical outcomes and treatment outcomes preceding Migalastat therapy. |
| | Secondary objectives |
| | To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment. |
| | To describe FACEs in accordance with different genoand phenotypic groups. |
| | To investigate the incidence and time to a first fatal or non-fatal cardiac, renal and cerebrovascular clinical event, separated by each category. |
| Country(-ies) of study | Denmark |

## STATEMENT OF COMPLIANCE

The study will be conducted in accordance with the Declaration of Helsinki principles, International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines, and applicable Danish regulations and laws. All personnel involved in the conduct of this study have completed human subjects' protection training.

## **SIGNATURE PAGE**

The signature below constitutes the approval of this protocol and the attachments and provides the necessary assurances that this study will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable regulations and guidelines.

| Principal I | nvestigator or Clinical Site Investigator: | |
|-------------|--------------------------------------------|-------|
| Signed: | | Date: |
| | Name: | |
| | Title: | |

## **Table of contents**

| Study information | 19 |
|---|---|
| Primary objectives | |
| Secondary objectives | 20 |
| STATEMENT OF COMPLIANCE | 21 |
| SIGNATURE PAGE | 22 |
| Table of contents | 23 |
| List of abbreviations | 25 |
| Responsible parties | 26 |
| Abstract | 28 |
| Primary outcomes | |
| Secondary outcomes | |
| Amendments and updates | |
| Milestones | |
| Rationale and background | |
| Research question and objectives | 32 |
| Research methods | 33 |
| Study design | |
| Endpoints | |
| Patient reported outcomes (PRO) | |
| Setting | |
| Study population | |
| Treatments | |
| Study workflow | |
| Variables | |
| Variables of interest at inclusion | |
| Exploratory outcome variables Other variables and exploratory outcome variables | |
| Safety variables | |
| Data sources | |
| Data sources for primary endpoints | |
| Other data sources | |
| Study size | |
| Data management | |
| Data collection | |
| Validation procedures | |
| Data management | |
| Medical coding | 45 |
| Serious Adverse Events/Adverse Events Data Reconciliation | 45 |
| Database lock | 45 |

| Data analysis | 45 |
|---------------------------------------------------------------------|----|
| Descriptive statistics | 45 |
| Handling of missing data | 46 |
| Primary endpoints analysis | 46 |
| Secondary endpoints analysis | 46 |
| Quality control | |
| Monitoring | 46 |
| Investigator training | 46 |
| Audits | |
| Inspections | |
| Limitations of the research methodology | 47 |
| Protection of human subjects | 47 |
| Ethics and Good Clinical Practice | 47 |
| Regulatory framework of the study | 47 |
| Independent Ethics Committee / Institutional Review Board | 47 |
| Subject information and consent | 47 |
| Subjects and data confidentiality | 47 |
| Subject Confidentiality | 47 |
| Data Confidentiality | 48 |
| Data handling and record keeping | |
| Record keeping and archiving | 48 |
| Transfer of Essential Documents | |
| Financing and insurance | |
| Financing | 48 |
| Management and reporting of adverse events/adverse reactions | 49 |
| Adverse event (AE) | 49 |
| Plans for disseminating and communicating study results | 49 |
| References | 50 |
| Annex 1. List of stand-alone documents | 52 |
| Annex 2. ENCePP checklist for study protocols | 52 |
| Annex 3. Additional information | |
| List annex 1.1 Description of participating clinical scientists and | |
| research staff | 53 |

## List of abbreviations

α-Gal A Alpha Galactosidase A

ACE Angiotensin-Converting Enzyme
ARB Angiotensin-Receptor Blockers

BPI Brief Pain Inventory

CRA Clinical Research Assistant

CRO Contract Research Organization
eCRF electronic Case Report Form
EDC Electronic Data Capture

ERT Enzyme Replacement therapy

ESRD End-Stage Renal Disease

FACE Fabry Associated Clinical Event

FPI First Patient In

GL-3/Gb3 Globotriaosylceramide Lyso Gb3 Globotriaosylsphingosine GCP Good Clinical Practices

GLA Galactosidase A
IgG Immunoglobulin G
LPO Last Patient Out
LV Left Ventricle

LVH Left Ventricular Hypertrophy
LVMI Left Ventricular Mass Index

MedDRA Medical Dictionary for Regulatory Activities

MSSI Mainz Severity Score Index

PBI Patient Benefit Index

PBQ Patient Benefit Questionnaire
PCA Principal Component Analysis

PI Principal Investigator

PNQ Patient Needs Questionnaire

PT Preferred Term
Q1 First Quartile
Q3 Third Quartile

SF-36v2 The Short Form (36) Health Survey version 2

SIV Site Initiation Visit

SmPC Summary of Product Characteristics

SOC System Organ Class

TSQM-9 Treatment Satisfaction Questionnaire for Medication v.9

QoL Quality of Life

SAE Serious Adverse Event

## **Responsible parties**

## **SPONSOR CONTACT DETAILS**

| Name | Rigshospitalet and Copenhagen University Department of Medical Endocrinology and Metabolism |
|---|---|
| Address | Rigshospitalet, Copenhagen University Hospital Blegdamsvej 9 DK-2100 Copenhagen Denmark |
| Phone number | +45 3545 2337 |

| COORDINATING INVESTIGATOR | |
|---|---|
| Name / Title | MD, PhD, Caroline Kistorp, Professor, Senior Consultant at Department of Medical Endocrinology and Metabolism, Rigshospitalet and Copenhagen University |
| Address | Rigshospitalet, Copenhagen University Hospital |
| | Blegdamsvej 9 |
| | DK-2100 Copenhagen |
| | Denmark |
| Phone/Fax | +45 22475699 |
| Email | caroline.michaela.kistorp@regionh.dk |

## **CONTRACT RESEARCH ORGANIZATIONS INFORMATION**

| Name | NOT APPLICABLE |
|---------|----------------|
| Address | |

| Phone/Fax |
|-----------|
| Email |

Participating clinical scientists and research staff will be described in Annex 1

## **Abstract**

| Title | Real World Evidence study of Danish Fabry patients: a > 20-year longitudinal retrospective analysis of prospectively collected data. |
|---|---|
| Rationale and background | Fabry is a rare X-linked metabolic lysosomal disorder caused by deficiency in the enzyme a-galactosidase A ( $\alpha$ -Gal A) by mutations in the <i>GLA</i> gene, encoding the $\alpha$ -Gal A enzyme, which catalyses glycosphingolipids, namely globotriaosylceramide (Gb3). Reduced or absent $\alpha$ -Gal A activity leads to accumulation of Gb3 in various organs as well as cellular dysfunction and inflammation causing phsyical symptoms and eventual organ failure. Migalastat, an oral chaperone therapy was approved for Fabry patients in 2016 providing an alternative to infusions with enzyme replacement every 2 weeks. Although the initial trials of Migalastat had some both short and extended outcome treatment comparisons, the overall evidence of clinical efficacy is based on too small numbers considering the heterogeneity of the Fabry patient population as well as the very slow progression of the disease. Though the body of real-world evidence is growing, there is a need for more publications of real-world long-term data on clinical outcomes with a focus on treatment with Migalastat. |
| | Research Question Is the incidence and prevalence of Fabry associated clinical events (FACEs) (cardiac, renal, and cerebrovascular) associated with sex, genotype, phenotype at time of diagnosis, biomarkers, and Fabry specific therapy? |
| | Objectives To investigate time to first Fabry associated clinical events (FACE) (cardiac, renal, and cerebrovascular) with particular focus on Migalastat clinical outcomes and treatment outcomes preceding Migalastat therapy. |
| Research question and objectives | To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment. |
| | To describe FACEs in accordance with different geno- and phenotypic groups. |
| | To investigate the incidence and time to a first fatal or non-fatal cardiac, renal, and cerebrovascular clinical event, separated by each category. |
| | Primary outcomes |
| | Time to first FACE (cardiac, renal, and cerebrovascular) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy. |

| | Secondary outcomes |
|---|---|
| | To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment. |
| | To describe FACEs in accordance with different geno- and phenotypic groups |
| | To investigate the incidence and time to a first fatal or non-fatal cardiac, renal and cerebrovascular clinical event, separated by each category. |
| Study design | Retrospective observational, single-center study from the Danish National Fabry Center. Describing treatment related outcomes in Fabry Disease over time. |
| Population | <ul> <li>Male and female patients with a diagnosis of Fabry Disease.</li> <li>Registred at the Danish National Fabry center, Rigshospitalet,<br/>Denmark from 01.01.2001.</li> </ul> |
| Variables | The primary endpoint is time to first FACE (cardiac, renal, or cerebrovascular events) since each baseline, with particular focus on the added value of the recent addition of Migalastat as a treatment option. Secondary endpoints are prevalence and incidence of FACEs and time to first FACE. Exploratory endpoints: Organ-specific biomarkers across modalities (auditory, lung, heart, kidney, skin, and neurological), and patient-reported outcomes evaluated by questionnaires. |
| Data sources | Electronic medical records and paper records. |
| Study size | Estimated 115 patients, which constitute all patients with a genetically verified diagnosis of Fabry disease in Denmark. |
| Data analysis | Primary endpoint will be addressed using event-driven statistics from a baseline based on the date of diagnosis and treatment initiation. Secondary analyses will address the individual parameters of the FACEs. Exploratory endpoints will rely on repeated measures statistical models to investigate the change in organ-specific function during the 20-year follow-up. Detailed description is found in statistical analysis plan (SAP). |
| Milestones | |
| Ethics Committee<br>Approval | Q3 2023 |
| Start of data collection | Q3 2023 |
| End of data collection | Q1 2024 |
| Study progress report | Q1 2024 |
| Interim report<br>(baseline data) | Q2 2024 |

| Registration in the EU<br>PAS register | Q3-4 2023 |
|----------------------------------------|-----------|
| Final report of study results | Q3 2024 |

## **Amendments and updates**

None

## **Milestones**

| Milestone | |
|-------------------------------------|-----------|
| Ethics Committee Approval | Q3 2023 |
| Start of data collection | Q3 2023 |
| End of data collection | Q1 2024 |
| Study progress report | Q1 2024 |
| Interim report (baseline data) | Q2 2024 |
| Registration in the EU PAS register | Q3-4 2023 |
| Final report of study results | Q3 2024 |

## Rationale and background

Fabry disease is a rare X-linked lysosomal disorder in lysosomes, resulting in a multisystemic disorder caused by deficiency in the enzyme  $\alpha$ -galactosidase A ( $\alpha$ -Gal A) due to mutations in the GLA gene, encoding the hydrolase  $\alpha$ -Gal A enzyme, which catalyses glycosphingolipids namely globotriaosylceramide (Gb3). Reduced or absent  $\alpha$ -Gal A activity leads to accumulation of Gb3 in the lysosomes of various organs, as well as cellular dysfunction and inflammation causing physical symptoms and eventual organ failure (1,2). Fabry disease as an X-linked disorder with a high penetrance, though not 100% in female heterozygotes, although the disease affects both males and females. With the X-linked nature, Fabry disease is suitable for an efficient, high diagnostic yield cascade screening over at least three generations surrounding an index-patient. The Danish National Fabry Centre has now more than 20 years of experience of cascade screening, which has provided a patient population of 115 male and female patients. The prevalence of Fabry disease in the Danish population is estimated to be 1:58000 (males 1:85000, females 1:44000) (3).

Primarily male patients, with early onset classical phenotypes have none or very low  $\alpha$ -Gal A activity, and they inevitably develop multiorgan failure without treatment (4). Patients with late onset of Fabry disease represent both males and females with higher  $\alpha$ -Gal A activity and variable degrees of organ involvement (5). Fabry disease can cause irreversible damage to multiple organs resulting in Fabry associated clinical events (FACEs) such as renal, cardiac, cerebrovascular events, and death (5).

The primary Fabry specific therapy has historically been enzyme replacement therapy (ERT), and as of 2016 an oral chaperone therapy, Migalastat, has been available, providing an alternative to ERT for patients with amenable mutations by increasing their endogenous  $\alpha$ -Gal A enzyme activity (6–14). However, real-world long-term data from well-characterised cohorts with available detailed clinical consecutive observations with focus on treatment with Migalastat and Fabry associated events has not been fully investigated (12–14).

## Research question and objectives

#### Research question

Is the incidence and prevalence of Fabry associated clinical events (FACEs) (cardiac, renal, and cerebrovascular) associated with sex, genotype, phenotype at time of diagnosis, biomarkers, and Fabry specific therapy?

#### **Objectives**

To investigate time to first Fabry associated clinical events (FACE) (cardiac, renal, and cerebrovascular) with particular focus on Migalastat clinical outcomes and treatment outcomes preceding Migalastat therapy.

To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment.

To describe FACEs in accordance with different geno- and phenotypic groups.

To investigate the incidence and time to a first fatal or non-fatal cardiac, renal and cerebrovascular clinical event, separated by each category.

#### **Primary objective**

To investigate time to first Fabry associated clinical events (FACEs) (cardiac, renal, and cerebrovascular) with particular focus on Migalastat clinical outcomes and treatment outcomes preceding Migalastat therapy.

#### **Secondary objectives**

To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment.

To describe FACEs in accordance with different geno- and phenotypic groups.

To investigate the incidence and time to a first fatal or non-fatal cardiac, renal and cerebrovascular clinical event, separated by each category.

#### **Exploratory objectives**

To describe disease progression with focus on organ involvement.

#### Research methods

#### Study design

Observational, retrospective, single-center study originating from the Danish National Fabry Centre, Centre of Cancer and Organ Disease, Department of Medical Endocrinology, Copenhagen University Hospital, Rigshospitalet. Patients are enrolled at the time of sampling leading to a genetically verified diagnosis of Fabry disease. Patients are followed from the day of enrolment until 31st of December 2022, having received yearly or bi-yearly evaluation during follow-up.

#### Method

Retrospective study of prospectively collected patient data with use of secondary patient data from both paper and electronic patient files. All patients are treatment naïve at time of diagnosis, which is defined as time point for a verified Fabry associated genetic mutation in the GLA gene. A baseline time point is further defined by switch of Fabry specific treatment. Both Migalastat and ERT will be studied retrospectively. Also untreated patients will be studied by assessment of relevant clinical and laboratory variables. The patients have been followed from 01.01.2001 until

31.12.2022. All patients with Fabry disease both receiving specific Fabry medication and untreated patients have been offered assessment yearly or every other year by thorough workup, including targeted examinations of organ function and symptoms known to be associated with Fabry Disease.

## **Endpoints**

#### **Primary endpoints**

The primary endpoint is time to first FACE (cardiac, renal, or cerebrovascular events) since each baseline, with particular focus on the added value of the recent addition of Migalastat as a treatment option.

FACEs are defined as the following:

- Cardiac clinical events:
  - Myocardial infarction
  - New symptomatic arrhythmia requiring medication, direct current cardioversion, or interventional procedure (e.g., ablation, pacemaker, or defibrillator implantation)
  - Unstable angina defined by national practice guidelines and accompanied by electrocardiographic changes and non-
  - Congestive heart failure requiring hospitalization
  - Any major cardiac medical procedure (e.g., valve replacement, stent-implantation, transplant or persistent atrial fibrillation)

ST segment elevation myocardial infarction [UA/NSTEMI]) and accompanied by electrocardiographic changes

- Cerebrovascular clinical events
  - Stroke (documented by a physician)
  - Transient ischemic attack (documented by a physician)
- Renal clinical events
  - Doubling of serum creatinine level from the start of analysis (2 consecutive values)
  - End-stage renal disease (ESRD) requiring long-term dialysis or transplantation
- Death due to FACEs

All FACEs will be analyzed together as a composite endpoint and separately in each category (cardiac, cerebrovascular, and renal).

## **Secondary endpoints**

The secondary endpoints

- The prevalence of FACEs from each baseline (diagnosis, and start of treatment) to compare between Migalastat-treated, ERT-treated patients and non-treated patients
- The incidence of FACEs from each baseline (diagnosis, and start of treatment) to compare between Migalastat-treated, ERT-treated patients and non-treated patients

- Time to the first cardiac, cerebrovascular, and renal clinical event separately by each specific category (including death in these categories) from start of treatment or baseline
- Incidence of cardiac, cerebrovascular, and renal clinical events separately by each specific category (including death in these categories)
- Occurrence of cardiac, cerebrovascular, and renal clinical events separately by each specific category (including death in these categories)
- Annualized rate of change in eGFR based on the Chronic Kidney Disease Epidemiology Collaboration equation (eGFR<sub>CKD-EPI</sub>) over time to compare between Migalastat-treated, ERT, and untreated patients
- The prevalence and incidence of a clinically significant change in mGFR and/or eGFR
   (according to KDIGO guidelines rapid progression is defined as a sustained decline in
   eGFR of more than 5 ml/min/1.73 m2 /yr) from each baseline (diagnosis, and start of
   treatment) to compare between Migalastat-treated, ERT-treated patients and non treated pts
- The prevalence and incidence of micro (> 30 mg/g creatinine) or macroalbuminuria (> 300) by urinary albumin/creatinine ratio (ACR) or urinary 24 h protein excretion from each baseline (diagnosis, and start of treatment) to compare between Migalastattreated, ERT-treated patients and non-treated pts

## **Exploratory organ specific Endpoints**

Reflecting the programme of the annual clinical examinations and questionnaires of the Danish Fabry patients.

**Lung capacity**: clinically significant changes in spirometry measures of obstructive and restrictive lung function evaluate by body plethysmography

Forced expiratory volume after 1 second (FEV1)

A clinically relevant change is defined as 25% decrease from baseline or as incident volume of 20% below predicted value according to an age- and sexadjusted reference range.

Forced vital capacity (FVC)

A clinically relevant change is defined as 25% decrease from baseline or as incident volume of 20% below predicted value according to an age- and sexadjusted reference range.

#### Neurological, audiological assessments

Standardized sweat test (hypo, normo, hyperhidrosis), standard unit of measure: mg pr.
 30 minutes

#### Standardized tilt-test (Presence of orthostatism - yes/no)

- Heart rate variability (Age-dependent impaired vs not)
- Audiogram (Impaired vs. not)
- Autonomic nerve function (small fibre assessment))
- Presence of Fabry associated abnormalities by brain MRI

#### Ophthalmological and dermatological assessments

- Presence of cornea versiculata
- · Presence of angiokeratoma

#### Composite phenotypic score

Mainz Severity Score Index (Composite score)

#### **Cardiac function** (evaluated by echocardiography)

- Left ventricular mass index (LVMi)
- Left ventricular ejection fraction (LVEF)
- Fractional shortening
- Left ventricular end diastolic and systolic volumes
- Mid-wall fractional shortening (MWFS)
- Left ventricular wall thickness
- NT-proBNP and high sensitive Troponin T will be analysed from the Danish Fabry biobank.

#### **Renal function**

#### Laboratory parameters:

- serum creatinine
- urine creatinine
- urine protein
- urine albumin
- urine ACR
- measured glomerular filtration rate by 99Tc-DTPA or 51Cr-EDTA

#### Patient reported outcomes (PRO)

SF-36 Health Questionnaire (Composite score)

- NHP-Health Profile (Daily living questionnaire composite score)
- Major Depression Inventory (Becks Depression Index II Composite score)

#### **Pharmacodynamic Endpoints**

Pharmacodynamic endpoints will be assessed by evaluations comparing Migalastat-treated and untreated patients and/or Migalastat-treated and ERT-treated patients:

- Plasma lyso-Gb<sub>3</sub>
- WBC α-Gal A enzyme activity
- Urinary and plasma Gb3, lyso-Gb3, α-GAL A enzyme activity
- Neutralizing antibodies with ERT

#### **Evaluation tools**

Data extraction from electronic and paper medical records. No specific evaluation test or tool required.

#### Setting

#### Study population

All patients from the Danish National Fabry Centre will be included, estimating the inclusion of 115 individuals (sex ratio [female:male] – 2:1). Pre-specified subgroups includes: non-amenable/amenable to Migalastat, males/females.

#### **Inclusion criteria**

- Established diagnosis of Fabry Disease based on genetic testing and alpha Gal-A activity in males and females.
- Data from baseline visit and at least one follow-up visit.

#### **Exclusion criteria**

Absence of data from baseline visit.

#### **Treatments**

#### Study treatment

No treatment will be evaluated prospectively. However, patients will be grouped according to treatment received during the treatment period (Migalastat, enzyme-replacement therapy or no treatment).

Patients who are switched from one treatment to another will be grouped according to current treatment at the assessment time point (if possible, according to a new baseline before switching).

Details of this procedure will depend on available information and numbers and cannot be described until all patients data have been collected.

## Symptomatic therapies

Data on nonspecific Fabry therapy such as ace enzyme inhibitors (ACE-I), angiotension-II blockers (AT-II), anticoagulants, statin, antiarrhythmic therapy, asthma/bronchodilator therapy, antidepressive therapy, as well as use of analgesics and other important concomitant medication will be recorded.

#### Other measures

If possible, information on comorbidities at each treatment start and switch will be recorded.

#### Study workflow

Fabry patients entered the study at their baseline visit (first visit in the center) from 2001 with last follow-up December 2022. Patient data will be grouped for the whole duration of the defined study period, with individual datapoints registered at the specific date of event/measurement. Ideally the datapoints will be used according to their specific dates but may be aggregated according to availability. Details is further described in the statistical analysis plan.

#### **Variables**

**Primary outcome variables** (Form to be filled at untreated baseline and every change in treatment status: From untreated to treated or vice versa, from one treatment to another.

Registration of treatment

All patients included in the trial are considered treatment naïve at inclusion in the observational period (01.01.2001). Registration of initiation, change or cessation of treatment will follow the following structure:

| Date | Drug | Action* | Dose | Dose interval | Comment |
|--------|--------|---------------|-----------|---------------|-----------|
| (Date) | (Name) | (Categorical) | (Integer) | (Comment) | (Comment) |

<sup>\*</sup>Action is restricted to four levels: initiation, increase, decrease, cessation.

| Cardiac events | | |
|----------------|--------------------------|--------|
| Date of event | Cardiac event | Yes/No |
| | Myocardial infarction | Yes |
| | | No |
| | Unstable angina pectoris | Yes |

| | | No |
|----|---------------------------------------------------------------|-----|
| PC | CI / CABG | Yes |
| | | No |
| Н | leart Failure | Yes |
| | | No |
| Aı | rrhythmia | Yes |
| (N | New onset of symptomatic arrhythmia requiring anti-arrhythmic | No |
| N | Medication) | |
| Н | leart procedure (pacemaker/ICD/valve surgery) | Yes |
| | | No |

| Renal events | | |
|---------------|--------------------------|--------|
| Date of event | Renal event | Yes/No |
| | Doubling of s-creatinine | Yes |
| | | No |
| | ESKD | Yes |
| | | No |

| Cerebrovascular events | | |
|------------------------|--------|-----|
| Date of event | Yes/No | |
| | Stroke | Yes |
| | | No |
| | TIA | Yes |
| | | No |

## Variables of interest at inclusion

Variables of interest at inclusion consists primarily of time invariant variables.

## <u>Demographics</u>

| Date of Birth | DDMMYYYY |
|---------------|-------------------------|
| Sex | Male Female |
| Ethnicity | White<br>Black<br>Asian |

| | Others |
|------|----------------|
| City | Residence City |

## Fabry-specific disease background

| A so of first supportance | Vacus |
|-------------------------------------|--------------------------|
| Age of first symptoms | Years |
| | <u> </u> |
| Age of diagnosis | Years |
| Fabry family history | Yes |
| | No |
| | Unknown |
| Index case | Yes |
| | No |
| ALPHA GAL ACTIVITY (LEUCO ASSAY) at | % of normal activity |
| inclusion | , |
| merasion | |
| MOLECULAR TEST | Amenable mutation found: |
| | Other mutations |
| 1 | other matations |

## **Exploratory outcome variables**

Variables concerning clinical presentation

| | Yes<br>No |
|---------------------|-----------|
| ANGIOKERATOMA | |
| CORNEA VERTICILLATA | Yes<br>No |
| ABDOMINAL PAIN | Yes<br>No |
| REFLUX | Yes<br>No |
| INDIGESTION | Yes<br>No |
| DIARRHEA | Yes<br>No |
| CONSTIPATION | Yes<br>No |
| DYSPNOEA | Yes<br>No |

| NEUROPATHIC PAIN | <ul><li>Yes</li><li>No</li></ul> |
|---------------------|----------------------------------|
| ACROPARAESTHAESIA | <ul><li>Yes</li><li>No</li></ul> |
| DEPRESSION SYMPTOMS | <ul><li>Yes</li><li>No</li></ul> |

Variables concerning organ dysfunction

| Lung capacity | |
|-------------------------------------------------|-----|
| Clinically significant Changes in spirometry of | Yes |
| obstructive function | No |
| Clinically significant changes in spirometry of | Yes |
| restrictive function | No |
| Neurological / Audiological | |
| Pathological heart rate variability | Yes |
| | No |

| Impaired hearing audiogram | Yes |
|----------------------------|-----|
| | No |
| Vertigo | Yes |
| | No |

| BLOOD PRESSURE | mmHg |
|----------------|------|
| Heart Rate | ВРМ |

| BUN | mmol/I |
|---|---|
| Plasma CREATININE | mmol/l |
| URINARY CREATININE | mg/dl |
| ALBUMIN/CREATININE RATIO | mg/g |
| PROTEINURIA | mg |
| GFR CKD-EPI | ml/min/1,73m <sup>2</sup> |
| mGFR | ml/min |
| Plasma Gb3 | microgram/ml |
| Plasma lysoGb3 | ng/ml |
| Urine GB3 | microgram/mmol creatinine |
| Alpha GAL-A activity (DBS or Leuco assay) | % normal activity and quantitative concentration (Method reference) |

## Variables concerning concomitant medication

The included concomitant medication to be recorded is restricted to medications believed to be of clinical interest. Medication will be recorded as to their use at inclusion and regarding their change throughout the study if possible.

| Concomitant medicati | on at inclusion |
|----------------------|-----------------|
| ACE-I/ ARB | Yes |
| | No |
| Beta-blocker | Yes |
| | No |
| Ca-blockers | Yes |
| | No |

| Diuretics | Yes |
|-----------|-----|
| | No |
| Statins | Yes |
| | No |

| Date | Drug | Action* | Dose | Dose interval | Comment |
|--------|--------|---------------|-----------|---------------|-----------|
| (Date) | (Name) | (Categorical) | (Integer) | (Comment) | (Comment) |

<sup>\*</sup>Action is restricted to four levels: Initiation, decrease, increase, cessation.

#### Other variables and exploratory outcome variables

## Safety variables

## **Safety Endpoints**

Although the study collects retrospective secondary data, adverse event reporting will be conducted, if necessary, in line with the requirements of each study supporter.

- SAEs
- Vital signs:
- resting systolic blood pressure
  - resting diastolic blood pressure
- Body weight
- Overall survival among all patients enrolled, as assessed by recorded patient deaths from any cause
- Laboratory parameters:
- serum creatinine
  - urine creatinine
  - urine protein
  - urine albumin
  - urine ACR
- ECGs
- ECHOs, including left ventricular mass index (LVMi), if medically indicated and requested by a physician
- Occurrence of male infertility.
- Infusion related reactions and other key safety events

#### Data sources

#### **Data sources for primary endpoints**

Electronic medical records, paper records and national medical records

#### Other data sources

Not applicable

#### Study size

The study is estimated to comprise of approximately 115 individuals with genetically verified Fabry Disease (Ratio of sex [female:male] 2:1).

#### Data management

#### **Data collection**

Investigators or other designated site staff are implemented in the project group will be trained in the specific procedural steps of the protocol, data extraction.

Study variables will be recorded in an electronic database/ CRF using validated and secure database in RedCap©. Patient data will be handled while preserving confidentiality. Investigators, or other designated site staff, will analyze all Fabry patients irrespective of disease-causing mutation and will extract clinical and laboratory parameters from original medical records (primary data sources).

## **Validation procedures**

A 10% random sample of records will be reviewed by a second independent observer to assure quality. The investigator team will discuss and resolve any noted discrepancies.

#### Case report form

All CRFs will be completed by the Investigators or other designated site staff who have been trained to record relevant information.

Data will be acquired retrospectively from medical documentation of enrolled patients.

Study variables will be recorded in a CRF designed for the specific purpose of this study. CRF design will be reviewed. At the end of data acquisition, the extent of missing values will be evaluated, and handled according to the description in the statistical analysis plan.

All patient data will be handled while preserving confidentiality.

#### **Data management**

All CRFs will be completed by the Investigators or other designated site staff who have been trained to record relevant information. Designated staff responsible for data acquisition should have higher medical education.

Data will be captured retrospectively from medical record documentation.

Study variables will be recorded in an electronic CRF by RedCap. CRFs will be reviewed for completeness at the end of document completion for data check (of missing data and/or specific questions requiring the investigators patient knowledge). All patient data will be handled preserving confidentiality.

#### Medical coding

Not applicable.

## Serious Adverse Events/Adverse Events Data Reconciliation

Although the study collects retrospective secondary data, reporting of adverse events will be conducted, if necessary, in line with the requirements of each study supporter. In the event of not previously reported serious adverse events or suspected, unexpected serious adverse reactions to a subscriber's product, these events will be reported to Competent Authorities within 24 hours.

#### **Database lock**

At the completion of data acquisition, all interested parties will be informed of impending data lock. Data lock will transpire if all parties agree, but before the independent validation by an external party and before statistical analysis.

#### Data analysis

#### **Descriptive statistics**

Analyses will be performed by descriptive statistical methods. Continuous variables will be described with number of patients with valid/missing observations, mean, standard deviation, median, minimum and maximum. Non-normally distributed data will be presented as median and interquartile range as appropriate. Categorical variables will be described by frequencies and related percentages. In addition to descriptive analysis, many of the endpoints will undergo statistical testing (i.e., p-values, confidence limits) to provide inferential summaries of subgroup comparisons (such as gender, age, ethnicity).

Details are going to be described in the Statistical Analysis Plan (SAP).

Analysis will be stratified by sex, age (> or <40 years), Fabry specific therapy (ERT treated (agalsidase alfa and beta separately), Migalastat treated, treatment naïve), baseline organ involvement (cardiac, renal, cerebrovascular, peripheral nervous system, and gastrointestinal system). Additional analysis may be required and carried out based on the results of the analyses mentioned above.

#### Handling of missing data

Missing data will not be imputed.

#### **Primary endpoints analysis**

Kaplan-Meier plots will be used to assess time to first Fabry associated clinical event (FACEs). Cox proportional hazard models will be used to assess the association between baseline characteristics and incident Fabry associated clinical event. The following baseline variables will be used in the model as covariables: age, time since diagnosis of Fabry disease, previous FACE (renal, cardiac, or cerebrovascular).

#### Patient benefit index

Not applicable

## Secondary endpoints analysis

Incidence rate of Fabry associated clinical events will be evaluated as events per 1000 patient – years

If data allows incidence and prevalence will be analyzed in subgroups (i.e., classic males, females, late-onset males, and females)

Renal, cerebrovascular, and cardiac function analyses will be performed in the same subgroups, as well as safety analyses per subgroup.

#### Quality control

#### **Monitoring**

#### **Investigator training**

Documents to perform the study will be mailed to physicians who agreed to participate, including the investigator agreements (fees agreement and confidentiality agreement).

Investigators and other designated site staff who have agreed to participate will be trained about the protocol, study procedures and CRF completion by teleconference or on-site visits.

Study variables will be recorded in a CRF, and patient data will be handled preserving confidentiality. Investigators, or other designated site staff will analyze all Fabry patients with amenable mutations and will extract clinical and laboratory features from original medical records (primary source).

#### **Audits**

Not applicable

#### **Inspections**

Not applicable

#### Limitations of the research methodology

The participating center has been selected as the Danish national Fabry center, with more than 20 years of experience managing patients with Fabry disease.

As the clinical data will be collected retrospectively, it is expected that some clinical data will be missing.

## **Protection of human subjects**

#### **Ethics and Good Clinical Practice**

The study will be conducted in accordance with ICH GCP. All applicable subject privacy requirements, and the ethical principles that are outlined in the Declaration of Helsinki 2013, including, but not limited to: Danish legal and health authorities and Ethical committee's review and favourable approval of study protocol and any subsequent amendments. The study will be reviewed and approved by the Danish Data Protection Agency, and the Danish Health Data Authority. With special regards to enrolment of patients who is dead, the study will be reviewed and approved by the Scientific Ethics Committee, The Capital Region, Denmark according to the specific legal requirements. Data will be anonymized (coded) when entered in the database.

#### Regulatory framework of the study

No drug will be evaluated prospectively, therefore, regulatory submission to the Danish Medical Association is not required in Denmark. Regarding data-collection, approval will be acquired from the legal regulatory authorities of the Capital Region of Denmark (see above).

#### **Independent Ethics Committee / Institutional Review Board**

No other Institute Review Board.

#### **Subject information and consent**

All patients will have provided written informed consent. The Study Team must maintain the original, signed Informed Consent/Assent Form. A copy of the signed Informed Consent/Assent Form must be given to the patient and/or their legally authorized representative.

A dated entry will be available in the patient's chart to confirm that informed consent/assent was obtained prior to any extraction of data and that the patient or their legally authorized representative received a copy of the signed informed consent/assent.

#### Subjects and data confidentiality

#### **Subject Confidentiality**

Information on patients' identity shall be considered as confidential for all effects and purposes. The patients' identity should not be revealed nor published under any circumstances. Patient data recorded in the CRF will be documented anonymously, coded with a patient number in such a way that only the investigator and site staff may associate data with an identified or identifiable

individual or his/her medical record. All other parties involved in data management, analysis and storage will receive, and subsequently analyze, non-identifiable patient data.

#### **Data Confidentiality**

By signing the investigator's confidentiality agreement, the investigator affirms to Amicus that information furnished by Amicus to the investigator will be kept in confidence and such information will be divulged to any expert committee, affiliated institution, and employees only under an appropriate understanding of confidentiality with such committee, affiliated institution, and employees.

#### Data handling and record keeping

By signing the investigator's confidentiality agreement, the investigator agrees that, within local regulatory restrictions and ethical considerations, Amicus or any Regulatory Agency may consult and/or copy study documents to verify the included data.

#### Record keeping and archiving

According to Danish law and to Amicus policies.

The investigator will keep a separate log of subjects' unique identification numbers in a tracker.

Only authorized persons will have access to identifiable personal details, if required for data verification. Data protection and privacy regulations will be observed in capturing, forwarding, processing, and storing subject data. If applicable, subjects will be informed accordingly and will be requested to give their consent on data handling procedures in accordance with national regulations.

In any presentations or in publications of the results of the study, the patients' identities will remain anonymous and confidential. Investigators, or investigator partners defined in annex 1 if applicable and various government health agencies may inspect the records of the study. Every effort will be made to keep the patients' personal medical data confidential.

During the development and analysis of the study, statistical program codes will be locally stored as documents according to best practices. Data protection laws in Denmark will be adhered to at all times. Further, the log file produced during the final run of each program will be stored locally at the investigator site as accompanying documents along with the results.

#### **Transfer of Essential Documents**

Not applicable

#### Financing and insurance

#### **Financing**

Senior researchers 2x50% data management 700,000 DKK

Specialist nurse to extract patient data 390,000 DKK

2 Medical students to extract data and manage data files 240,000 DKK

Meetings, IT access, literature review, publication costs 70,000 DKK

#### Total 1,400,000 DKK

Amicus sponsored

#### **Insurance**

Not applicable

# Management and reporting of adverse events/adverse reactions

#### Adverse event (AE)

Collection of adverse events as Individual Case Safety Reports (ICSRs) is not required from such retrospective analyses of patient medical records as it is secondary data.

#### Plans for disseminating and communicating study results

The study, and study results, will be disclosed on clinicaltrials.gov and other relevant clinical study disclosure websites in accordance with relevant AMICUS policies. The primary publication is expected to be in an internationally recognised journal, with the Scientific Committee forming the majority of the authorship. Thereafter, any secondary publications will reference the original publication and will be authored in accordance with International Committee of Medical Journal Editors (ICMJE) requirements.

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator is encouraged to share the summary results with the study subjects, as appropriate.

## References

- 1. Germain DP. Fabry disease. Orphanet J Rare Dis. 2010;5(1):30.
- 2. Sanchez-Nino MD, Sanz AB, Carrasco S, Saleem MA, Mathieson PW, Valdivielso JM, et al. Globotriaosylsphingosine actions on human glomerular podocytes: implications for Fabry nephropathy. Nephrol Dial Transplant. 2011 Jun 1;26(6):1797–802.
- 3. Effraimidis G, Rasmussen ÅK, Dunoe M, Hasholt LF, Wibrand F, Sorensen SS, et al. Systematic cascade screening in the Danish Fabry Disease Centre: 20 years of a national single-centre experience.

  Branchini A, editor. PLoS One. 2022 Nov 16;17(11):e0277767.
- Waldek S, Patel MR, Banikazemi M, Lemay R, Lee P. Life expectancy and cause of death in males and females with Fabry disease: Findings from the Fabry Registry. Genet Med [Internet]. 2009;11(11):790–6. Available from: https://doi.org/10.1097/GIM.0b013e3181bb05bb
- 5. Ortiz A, Germain DP, Desnick RJ, Politei J, Mauer M, Burlina A, et al. Fabry disease revisited: Management and treatment recommendations for adult patients. Mol Genet Metab. 2018 Apr;123(4):416–27.
- 6. Feldt-Rasmussen U, Hughes D, Sunder-Plassmann G, Shankar S, Nedd K, Olivotto I, et al. Long-term efficacy and safety of Migalastat treatment in Fabry disease: 30-month results from the open-label extension of the randomized, phase 3 ATTRACT study. Mol Genet Metab. 2020 Sep;131(1–2):219–28.
- 7. Schiffmann R, Bichet DG, Benjamin E, Wu X, Giugliani R. The Migalastat GLP-HEK assay is the gold standard for determining amenability in patients with Fabry disease. Mol Genet Metab Reports. 2019 Sep;20(July):100494.
- 8. Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, et al. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016;375(6):545–55.
- 9. Hughes DA, Nicholls K, Shankar SP, Sunder-Plassmann G, Koeller D, Nedd K, et al. Oral pharmacological chaperone Migalastat compared with enzyme replacement therapy in Fabry disease: 18-month results from the randomised phase III ATTRACT study. J Med Genet. 2017 Apr;54(4):288–96.
- 10. Schiffmann R, Bichet DG, Jovanovic A, Hughes DA, Giugliani R, Feldt-Rasmussen U, et al. Migalastat improves diarrhea in patients with Fabry disease: clinical-biomarker correlations from the phase 3 FACETS trial. Orphanet J Rare Dis. 2018 Dec 27;13(1):68.
- 11. Germain DP, Nicholls K, Giugliani R, Bichet DG, Hughes DA, Barisoni LM, et al. Efficacy of the pharmacologic chaperone Migalastat in a subset of male patients with the classic phenotype of Fabry disease and Migalastat-amenable variants: data from the phase 3 randomized, multicenter, double-blind clinical trial and extension study. Genet Med. 2019 Sep;21(9):1987–97.
- 12. Nowak A, Huynh-Do U, Krayenbuehl P, Beuschlein F, Schiffmann R, Barbey F. Fabry disease genotype, phenotype, and Migalastat amenability: Insights from a national cohort. J Inherit Metab Dis. 2020 Mar 30;43(2):326–33.
- 13. Riccio E, Zanfardino M, Ferreri L, Santoro C, Cocozza S, Capuano I, et al. Switch from enzyme replacement therapy to oral chaperone Migalastat for treating fabry disease: real-life data. Eur J Hum Genet. 2020 Dec 9;28(12):1662–8.
- 14. Müntze J, Gensler D, Maniuc O, Liu D, Cairns T, Oder D, et al. Oral Chaperone Therapy Migalastat for Treating Fabry Disease: Enzymatic Response and Serum Biomarker Changes After 1 Year. Clin

Pharmacol Ther. 2019 May 13;105(5):1224–33.

## Annex 1. List of stand-alone documents

Documents listed in Annex 1 can be maintained separately from the study protocol. They should be clearly identifiable and provided on request. Write "None" if there is no document or list documents in a table as indicated below.

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 1 | xx.xx.2023 | Text | Update | Description of participating clinical scientists and research staff |

## Annex 2. ENCePP checklist for study protocols

A copy of the ENCePP Checklist for Study protocols available at <a href="http://www.encepp.eu/standards">http://www.encepp.eu/standards</a> and guidances/index.html completed and signed by the main author of the study protocol should be included in Annex 2.

The checklist will facilitate the review of the protocol and evaluation of whether investigators have considered important methodological aspects.

In question 9.5 of the Checklist, Revision 1:

"Study start" means "Start of data collection"

## **Annex 3. Additional information**

Additional annexes may be included if necessary.

<sup>&</sup>quot;Study progress" means "Progress report(s)"

<sup>&</sup>quot;Study completion" means "End of data collection"

<sup>&</sup>quot;Reporting" means "Final report of the study results"

# **List annex 1.1** Description of participating clinical scientists and research staff

| DocuSian | Envelope I | D٠ | C59C9E98 | 700F | 4916 | -8D21 | -R23F | R6F | C.5 | SF |
|---|---|---|---|---|---|---|---|---|---|---|
| DUCUSIUII | LIIVEIODE I | <b>ப</b> . | COSCSESO | - / ບບ - | 4310 | -0021 | -DZJL | ப்பட | . UJ | $\omega_{\mathbf{L}}$ |

THIS FINAL PAGE IS BLANK.